CLINICAL TRIAL: NCT03766503
Title: Daily Delivery and Supervision of Psychotropic Medication for High-Risk Patients With Severe and Persistent Mental Illness
Brief Title: Daily Delivery and Supervision of Psychotropic Medication for High-Risk Patients With Severe/Persistent Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Winnipeg Regional Health Authority (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: H2016:321
Record Dates: First submitted 2018-05-03; First posted 2018-12-06 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Medication Adherence
Keywords: Medication adherence; Severe and persistent mental illness
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: The main study intervention is the daily witnessing of participants while they self-administer their medications by trained pharmacy staff to ensure compliance. The staff in question will be provided by Leila pharmacy and will in addition provide support so that individuals can transition back into living independently through reminders to attend regularly scheduled medical appointments and counseling on correct use of prescribed medications.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): The main study intervention is the daily witnessing of participants while they self-administer their medications by trained pharmacy staff to ensure compliance. The staff in question will be provided by Leila pharmacy and will in addition provide support so that individuals can transition back into living independently through reminders to attend regularly scheduled medical appointments and counseling on correct use of prescribed medications.
  Interventions: Other: Daily

INTERVENTIONS:
Other: Daily — The main study intervention is the daily witnessing of participants while they self-administer their medications by trained pharmacy staff to ensure compliance. The staff in question will be provided by Leila pharmacy and will in addition provide support so that individuals can transition back into living independently through reminders to attend regularly scheduled medical appointments and counseling on correct use of prescribed medications.

SUMMARY:
The main study intervention is the daily witnessing of participant self-administration of medications by trained pharmacy staff to ensure compliance. The staff in question will be provided by Leila pharmacy and will in addition provide support so that individuals can transition back into living independently through reminders to attend regularly scheduled medical appointments and counseling on correct use of prescribed medications.

DETAILED DESCRIPTION:
The program is designed to serve individuals with severe and persistent mental illnesses who have been repeatedly hospitalized, are repeat users of community crisis services, or are frequently in contact with the criminal justice system. There are several objectives of this new approach. First, the investigators believe that these patients are invested in working with the daily dispensing program to stay well, but individual factors related to their personal background or symptoms of their illness contribute to frequent non-adherence to medications. Non-adherence to medications then leads to behaviour that results in frequent use of very expensive services such as the criminal justice system, acute care hospital beds, and crisis services. Working collaboratively with the patient to improve adherence to medications in partnership with a private pharmacy that absorbs costs of the program is a less coercive model than injectable medications, which is the current standard for working with this population. In addition, oral medications are much less expensive than the newer injectable antipsychotics and the costs of running a "depot clinic" where the injectable medications are provided. At this time, there has been no effective program to ensure compliance with oral medications in the published literature.

The primary purpose of this study is to evaluate the effectiveness of this new model for decreasing the harmful effects of relapses to psychosis resulting from non-adherence to medications. Specifically, the investigators plan to examine whether or not this program results in less use of crisis services, acute care hospitalization and less contact with the criminal justice system. The investigators plan to evaluate client response through a self-reported measure and to assess client satisfaction by conducting participant satisfaction survey for the program. Key stakeholders will be engaged during the process (e.g., community mental health workers, probation officers, pharmacists) to gather information and suggestions regarding the daily dispensing program. Based on feedback from clients and stakeholders, the investigators will then aim to implement improvements to the process to optimize its effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Individuals currently enrolled in the new daily dispensing program
* Individuals with severe and persistent mental illnesses
* Individuals who have been repeatedly hospitalized, are repeat users of community crisis services, or are in frequently in contact with the criminal justice system
* Individuals who are involved in the Forensics program.

Exclusion Criteria:

* Individuals who are not currently in the Forensics program
* Individuals who are part of the daily dispensing program, but are not Forensic outpatients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-10-15 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-02-11 (Actual)

PRIMARY OUTCOMES:
Patient Self-Report Measure (Client Coercion Survey) | This study will employ a crossover design where data is collected for 12 months during the study and compared to baseline data retrieved for 12 months for each patient before enrollment into the project.
  The questionnaire asks about the client's perceptions of care which will help measure the effectiveness of the study's recovery intervention (Daily Dispensing program) by evaluating patient response to the program through this self-reported measure. The measure is composed of three subscales: Perceived Coercion (items scored as False=1; True/Don't Know=0); Negative Pressures (items scored as False=1; True/Don't Know=0; except item 12 is reverse scored); Voice (items scored as False=1; True/Don't Know=0; except item 13 which is reverse scored). The Perceived Coercion subscale ranges from 0 (minimum score) to 5 (maximum score) and lower values reflect better outcomes; the Negative Pressures subscale ranges from 0 (minimum score) to 6 (maximum score) and higher values reflect better outcomes; the Voice subscale ranges from 0 (minimum score) to 3 (maximum score) and lower values reflect better outcomes. The subscales will not be combined to compute a total score.

SECONDARY OUTCOMES:
Stakeholder survey | This study will employ a crossover design where data is collected for 12 months during the study and compared to baseline data retrieved for 12 months for each patient before enrollment into the project.
  The researchers will engage key stakeholders during the project (e.g., community mental health workers, psychiatrists, pharmacists) to gather information and suggestions regarding the Daily Dispensing program. Based on feedback stakeholders, the researchers will then aim to implement improvements to the program to optimize its effectiveness. The survey uses a 5 point Likert scale and items are scored from 1 to 5 (and the negative questions items 8, 10, 12 are reverse scored) with lower scores indicating better outcomes. The scale contains 11 items that can be summed (items: 3-12, 15) - the maximum score for this scale is 55 (5 x 11 items) and the minimum score is 11 (1 x 11 items). The Stakeholder Survey has no subscales. The survey also features 7 descriptive items (items: 1, 2, 13, 14, 16-19) and these will be reported.
Client Satisfaction Measure | This study will employ a crossover design where data is collected for 12 months during the study and compared to baseline data retrieved for 12 months for each patient before enrollment into the project.
  The survey measures clients' satisfaction regarding program and consists of several domains but no real subscales: accessibility, availability of resources, continuity of care, outcome of care, humanness of program staff, information gathering, information giving, pleasantness of surroundings, competence of staff, and quality of program. The survey was further modified by the Daily Dispensing team. The survey uses a 5 point Likert scale and items are scored from 1 to 5 with lower scores indicating better outcomes. There are no reverse scored items. The scale contains 26 items that can be summed - the maximum score for the Client Satisfaction Scale is 130 (5 x 26 items) and the minimum score is 26 (1 x 26 items). Items 27-29 are descriptive and these will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Waldman, MD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Canada

IPD SHARING:
Plan to Share IPD: Yes
All patient personal health information: Personal Health Information Number (PHIN), name and date of birth will be stored in a secured database (REDCAP) for the duration of the project. Analysis will be done on aggregate data only stripped from personal health identifiers. Database will be archived in REDCAP with access only by authorized individuals.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be collected over a span of 12 months and be retained for seven years.
Access Criteria: Only authorized project staff will have access to patient medical information. Aggregate data will be made available for sharing with other organizations.

REFERENCES:
- [Background] Emsley R, Oosthuizen P, Koen L, Niehaus D, Martinez L. Comparison of treatment response in second-episode versus first-episode schizophrenia. J Clin Psychopharmacol. 2013 Feb;33(1):80-3. doi: 10.1097/JCP.0b013e31827bfcc1. PMID 23277247
- [Background] Goeree R, Farahati F, Burke N, Blackhouse G, O'Reilly D, Pyne J, Tarride JE. The economic burden of schizophrenia in Canada in 2004. Curr Med Res Opin. 2005 Dec;21(12):2017-28. doi: 10.1185/030079905X75087. PMID 16368053
- [Background] Keers R, Ullrich S, Destavola BL, Coid JW. Association of violence with emergence of persecutory delusions in untreated schizophrenia. Am J Psychiatry. 2014 Mar;171(3):332-9. doi: 10.1176/appi.ajp.2013.13010134. PMID 24220644
- [Background] Patel MX, de Zoysa N, Bernadt M, Bindman J, David AS. Are depot antipsychotics more coercive than tablets? The patient's perspective. J Psychopharmacol. 2010 Oct;24(10):1483-9. doi: 10.1177/0269881109103133. Epub 2009 Mar 20. PMID 19304865
- [Background] Patel MX, de Zoysa N, Bernadt M, David AS. A cross-sectional study of patients' perspectives on adherence to antipsychotic medication: depot versus oral. J Clin Psychiatry. 2008 Oct;69(10):1548-56. doi: 10.4088/jcp.v69n1004. Epub 2008 Sep 23. PMID 19192437
- [Background] Rossler W, Salize HJ, van Os J, Riecher-Rossler A. Size of burden of schizophrenia and psychotic disorders. Eur Neuropsychopharmacol. 2005 Aug;15(4):399-409. doi: 10.1016/j.euroneuro.2005.04.009. PMID 15925493
- [Background] Schooler NR. Relapse prevention and recovery in the treatment of schizophrenia. J Clin Psychiatry. 2006;67 Suppl 5:19-23. PMID 16822093
- [Background] Thornicroft G, Brohan E, Rose D, Sartorius N, Leese M; INDIGO Study Group. Global pattern of experienced and anticipated discrimination against people with schizophrenia: a cross-sectional survey. Lancet. 2009 Jan 31;373(9661):408-15. doi: 10.1016/S0140-6736(08)61817-6. Epub 2009 Jan 21. PMID 19162314
- [Result] Angermeyer MC, Matschinger H. The stereotype of schizophrenia and its impact on discrimination against people with schizophrenia: results from a representative survey in Germany. Schizophr Bull. 2004;30(4):1049-61. doi: 10.1093/oxfordjournals.schbul.a007120. PMID 15954207

DOCUMENTS (2):
  • Study Protocol (2018-01-17): https://cdn.clinicaltrials.gov/large-docs/03/NCT03766503/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-17): https://cdn.clinicaltrials.gov/large-docs/03/NCT03766503/SAP_001.pdf